CLINICAL TRIAL: NCT06356792
Title: The Associations Between History of Recurrent Miscarriage and Obstetric and Perinatal Outcomes in the Subsequent Pregnancy
Brief Title: Obstetrics , Prenatal Outcomes in Recurrent Miscarriage
Acronym: OBPORPL
Status: Recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Reem Salah Abdelkareem Ahmed, Principal investigator, Assiut University
Other Study IDs: Obstetrics outcome in Abortion
Record Dates: First submitted 2024-03-21; First posted 2024-04-10 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Recurrent Miscarriage
MeSH Terms: conditions — Abortion, Habitual

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The effect of recurrent miscarriage on the outcome of the current pregnancy and if there's a relation between it and adverse out come

ELIGIBILITY:
Inclusion Criteria:

1- patients who had ≥2 abortions during early pregnancy 2.patients had no abnormal reproductive tract anatomy 3. Pregnant in single fetus

Exclusion criteria:

chronic hypertension, chronic kidney diseases autoimmune diseases multiple pregnancy

Min Age: 17 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: patients who had ≥2 abortions during early pregnancy, patients had no abnormal reproductive tract anatomy , single fetus
Sampling Method: Non-Probability Sample
Enrollment: 102 (Estimated)
Dates: Start 2024-04-21 (Estimated); Primary Completion 2025-03-21 (Estimated); Study Completion 2025-03-21 (Estimated)

PRIMARY OUTCOMES:
If there's relation between recurrent abortion and having a medical disorder during current pregnancy | 2023 to 2025

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University, Asyut, Egypt